CLINICAL TRIAL: NCT00454168
Title: A Phase 3, Randomized, Double-Blind, Multicenter Study of Proteinase 3 PR1 Peptide Mixed With Montanide ISA-51 VG Adjuvant and Administered With GM-CSF in Elderly Patients With AML in First Complete Remission or Adults in Second Complete Remission: A Pivotal Study
Brief Title: Vaccine Therapy and GM-CSF in Treating Patients With Acute Myeloid Leukemia in Remission
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Vaccine Company (Industry)
Responsible Party: Regulatory Protocol Associate, Vaccine Company
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000510853; VACCINE-PR1-104; UCCRC-14613B
Record Dates: First submitted 2007-03-27; First posted 2007-03-30 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2009-02

CONDITIONS: Leukemia
Keywords: adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myelomonocytic leukemia (M4); adult acute promyelocytic leukemia (M3); secondary acute myeloid leukemia; adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — sargramostim

ARMS (2):
- Arm I (Experimental): Patients receive PR1 leukemia peptide vaccine and sargramostim (GM-CSF) subcutaneously.
  Interventions: Biological: PR1 leukemia peptide vaccine; Biological: sargramostim
- Arm II (Active Comparator): Patients receive placebo vaccine and GM-CSF subcutaneously.
  Interventions: Biological: sargramostim; Other: placebo

INTERVENTIONS:
Biological: PR1 leukemia peptide vaccine — Given subcutaneously
  Arms: Arm I
Biological: sargramostim — Given subcutaneously
Other: placebo — Given subcutaneously
  Arms: Arm II

SUMMARY:
RATIONALE: Vaccines made from a peptide may help the body build an effective immune response to kill cancer cells. Colony-stimulating factors, such as GM-CSF, increase the number of white blood cells and platelets found in bone marrow or peripheral blood. Giving vaccine therapy together with GM-CSF may be an effective treatment for acute myeloid leukemia. It is not yet known whether giving vaccine therapy together with GM-CSF is more effective than giving placebo together with GM-CSF in treating acute myeloid leukemia.

PURPOSE: This randomized phase III trial is studying vaccine therapy and GM-CSF to see how well they work compared with a placebo and GM-CSF in treating patients with acute myeloid leukemia in remission.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare improvement of overall survival of patients with acute myeloid leukemia treated with PR1 leukemia peptide vaccine and sargramostim (GM-CSF) vs placebo vaccine and GM-CSF.

Secondary

* Compare improvement of relapse-free survival of patients treated with these regimens.
* Compare remission duration in patients treated with these regimens.
* Compare immune response, as measured by PR1-HLA-A2 tetramer assay, in patients treated with these regimens.

OUTLINE: This is a randomized, placebo-controlled, multicenter study. Patients are stratified according to age and complete remission (CR) (≥ 18 years of age and in second CR vs ≥ 55 years of age and in first CR), type of acute myeloid leukemia (de novo vs secondary), and cytogenetics (unfavorable vs favorable and intermediate). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive PR1 leukemia peptide vaccine and sargramostim (GM-CSF) subcutaneously (SC).
* Arm II: Patients receive placebo vaccine and GM-CSF SC.

PROJECTED ACCRUAL: A total of 244 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML), defined by the presence of > 20% blasts in marrow or blood, including the following subtypes:

  * De novo AML, defined as AML with no clinical history of prior myelodysplastic syndromes (MDS) or myeloproliferative disorder (MPD) or exposure to potentially leukemogenic therapies or agents
  * Secondary AML, defined as the following:

    * AML secondary to prior existing MDS or MPD or development of AML secondary to proven leukemogenic exposure
    * History of fatigue, bleeding, or recurrent infections preceding diagnosis of AML by ≥ 1 month with confirmation of existing peripheral blood film that demonstrates morphologic dysplasia
* In first complete remission (CR) (patients ≥ 55 years of age) OR second CR (patients ≥ 18 years of age) within the past month

  * FAB stages M0-M2 and M4-M7 allowed if in first CR

    * No acute promyelocytic leukemia in first CR
  * FAB stages M0-M7 allowed if in second CR
  * Marrow blast count < 5% (≤ 200 nucleated cell count)

    * No blasts in blood
* HLA-A2 positive at 1 allele
* No extramedullary disease
* No Auer rods
* No active meningeal or CNS leukemia

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy must not be severely limited by other diseases
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Bilirubin < 2 mg/mL
* ALT < 2 times upper limit of normal
* Creatinine ≤ 1.6 mg/mL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Antineutrophil cytoplasmic antibody negative
* No serious medical condition, laboratory abnormality, or psychiatric illness that would preclude study compliance or increase risk to patient
* No other malignancy within the past 5 years except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast
* No known allergy to incomplete Freund's adjuvant
* No hypercalcemia
* No progressive viral or bacterial infection

  * Must be afebrile for 7 days without antibiotics
* No symptomatic cardiac disease
* LVEF ≥ 40%
* No symptomatic pulmonary disease
* FEV_1, FVC, and DLCO ≥ 50% of predicated (without bronchodilator)
* No history of HIV positivity or AIDS
* No known hypersensitivity to sargramostim (GM-CSF), yeast-derived products, or any component of this product
* No history of Wegener's granulomatosis or vasculitis

PRIOR CONCURRENT THERAPY:

* Recovered from prior surgery and/or radiotherapy
* No prior allogeneic or syngeneic stem cell transplantation
* No prior solid organ transplantation
* No prior vaccine therapy for AML
* More than 28 days since prior chronic use (> 2 weeks) of corticosteroids > 10 mg/day (prednisone [or equivalent])

  * Concurrent topical or inhaled corticosteroids allowed
* More than 3 months since prior experimental therapy, cyclosporine, or tacrolimus
* No concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2005-05; Primary Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Relapse-free survival
Remission duration
Immune response as measured by PR1-HLA-A2 tetramer assay

CONTACTS AND LOCATIONS:
Overall Officials: Craig S. Rosenfeld, MD, Study Chair — The Vaccine Company
Locations (15):
- United States (15):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Vaccine Company, South San Francisco, California
  - Rush Cancer Institute at Rush University Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - St. Francis Hospital Cancer Care Services, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cancer Care Centers of South Texas - Southeast, San Antonio, Texas